CLINICAL TRIAL: NCT04707014
Title: Effectiveness of Hypnoanalgesia for Dermatological Surgery in Children: Randomised Clinical Trial
Brief Title: Hypnoanalgesia for Dermatological Surgery in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario de Toledo (Other)
Responsible Party: Principal Investigator, JUANA MARIA PELAEZ PEREZ, Anesthesiologist, Complejo Hospitalario de Toledo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHT00028
Record Dates: First submitted 2020-09-17; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia
Keywords: analgesia; anxiety; pain; paediatric surgery; dermatology; Hypnosis; Nervous System Diseases Central; Hypnotics and Sedatives; Nervous System Depressants; Physiological Effects of Drugs
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Pain; Central Nervous System Diseases | interventions — Hypnosis; Hypnosis, Anesthetic

STUDY DESIGN:
Intervention Model Description: Patients are randomly distributed to one of the following groups:
  Intervention group: Technique of rapid conversational hypnosis, with focus on therapeutic suggestion (guiding the patient into a hypnotic trance), adapted to child's cognitive development. Induction with hypnotic suggestion focuses and accompanies the child's body sensations and allows their active participation. After standard sedation, therapeutic suggestion is maintained throughout the surgery and in the post-hypnotic period before awakening.
  Control group: High-tech distraction technique (Apple®), passive and chosen by the child, either an animated video or his or her favourite music. After standard intravenous sedation, the child is taken to the operating theatre to watch his or her favourite video or music and this is maintained throughout the procedure.
Who Masked: Outcomes Assessor
Masking Description: Different investigators are assigned to each phase of the study, with one designated as responsible for recruitment (MQD), another for intervention and control (JMPP), and another for subsequent evaluation in the post-anaesthesia recovery unit (URPA) and at 24 hours (responsible nursing staff).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention-Distraction techniques (Placebo Comparator): A high-tech distraction technique (Apple®), passive and chosen by the child, either an animated video or his or her favourite music. After standard intravenous sedation, the child is taken to the operating theatre to watch his or her favourite video or music and this is maintained throughout the procedure.
  Interventions: Behavioral: Attention-distracting techniques
- HIPNOSIS GROUP (Experimental): A technique of rapid conversational hypnosis, with focus on therapeutic suggestion (guiding the patient into a hypnotic trance), adapted to the child's cognitive development. Induction with hypnotic suggestion focuses and accompanies the child's body sensations and allows their active participation. After standard sedation, therapeutic suggestion is maintained throughout the surgery and in the post-hypnotic period before awakening.
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — Rapid conversational hypnosis
  Other Names: Hypnoanalgesia; Hypnosedation
  Arms: HIPNOSIS GROUP
Behavioral: Attention-distracting techniques — i-pad with movies, games and music
  Arms: Attention-Distraction techniques

SUMMARY:
This randomized clinical trial will evaluate the effect of hypnosedation on the need of sedation and analgesia in a pediatric population undergoing dermatological surgery, both during the procedure, and 24 hours after surgery. In addition, a secondary objetive is to evaluate the effect by specific age groups.

DETAILED DESCRIPTION:
In this clinical trial, pediatric patients scheduled for removal of benign skin lesions in a single center willbe randomised to receive hypnosis (intervention group) or attention-distracting techniques (control group). Endpoints will be the sedative dose (propofol) during surgery, and the need for analgesia (paracetamol and others) immediately after surgery (recovery) and after 24 hours. Randomization will be systematic in blocks depending on the day the surgery is programmed. Hypnosis will be delivered by an experienced anesthesist trained in the technique. Patients and families will be informed of the special treatment during surgery, but will be unaware of whether the patients are experiencing distraction or hypnosis techniques. Distraction is already a useful technique, and it is expected that patients will be satisfied with the procedure; however, the hypothesis to be tested is that hypnosis reduces the need for sedation and analgesia compared to distraction techniques, as well as improves satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. A class I or II of anaesthetic risk according to the American Society of Anesthesiologists,
2. to be in a percentile between P3 and P97 in weight and height,
3. without known drug allergies, and
4. having fasted 6 hours for solids and 2 hours for water.

Exclusion Criteria:

1. Children with diagnosed mental retardation or attention deficit,
2. behavioural disorders,
3. previous treatment with hypnosis,
4. history of neurological pathology or psychomotor retardation,
5. previous pain-related pathology,
6. obstructive sleep apnoea syndrome (OSAS)

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Total dose of propofol in mg/kg | During surgery (Intra-operative)
  Measured in mg/kg weight
Total dose of propofol in mg | During surgery (Intra-operative)
  Measured in total mg
Additional need for opioids during surgery | During surgery (Intra-operative)
  Yes/no

SECONDARY OUTCOMES:
Pain intensity in older children post-operative | Immediately post-operative while on recovery unit
  0-10 visual analogue scale (VAS) administered by a blinded nurse, with higher values indicating higher levels of pain
Pain intensity in younger children post-operative | Immediately post-operative while on recovery unit
  0-10 Faces Pain Scale - Revised (FPS-r) administered by a blinded nurse, with higher values indicating higher levels of pain
Pain intensity in older children after 24 hours | 24 hours after discharge
  0-10 visual analogue scale (VAS) administered over the phone by a blinded nurse, with higher values indicating higher levels of pain
Pain intensity in younger children after 24 hours | 24 hours after discharge
  0-10 Faces Pain Scale - Revised (FPS-r) administered over the phone by a blinded nurse, with higher values indicating higher levels of pain
Analgesic need | 24 hours after discharge
  Recorded by a blinded nurse at reanimation unit as yes/no
Analgesic needs | 24 hours after discharge
  Recorded by a blinded nurse by telephone call as yes/no

OTHER OUTCOMES:
Degree of satisfaction with the procedure | 24 hours after discharge
  Validated survey with score 1-10 administered at the time of discharge to children and their guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Juana Maria PELAEZ PEREZ, PH, Principal Investigator — Complejo Hospitalario Toledo
Locations (1):
- Complejo Hospitalario Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Yes
Any document upon reasonable request to the PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Up to 1 year after publication
Access Criteria: Justified interest in data. By e-mail to PI

REFERENCES:
- [Background] Friedrichsdorf SJ, Kohen DP. Integration of hypnosis into pediatric palliative care. Ann Palliat Med. 2018 Jan;7(1):136-150. doi: 10.21037/apm.2017.05.02. Epub 2017 Jun 27. PMID 28866891
- [Background] Kendrick C, Sliwinski J, Yu Y, Johnson A, Fisher W, Kekecs Z, Elkins G. Hypnosis for Acute Procedural Pain: A Critical Review. Int J Clin Exp Hypn. 2016;64(1):75-115. doi: 10.1080/00207144.2015.1099405. PMID 26599994
- [Background] Brown ML, Rojas E, Gouda S. A Mind-Body Approach to Pediatric Pain Management. Children (Basel). 2017 Jun 20;4(6):50. doi: 10.3390/children4060050. PMID 28632194
- [Background] Friedrichsdorf SJ, Goubert L. Pediatric pain treatment and prevention for hospitalized children. Pain Rep. 2019 Dec 19;5(1):e804. doi: 10.1097/PR9.0000000000000804. eCollection 2020 Jan-Feb. PMID 32072099

DOCUMENTS (3):
  • Study Protocol: HYPNOANALGESIA IN PEDIATRIC DERMATOLOGICAL SURGERY (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04707014/Prot_000.pdf
  • Statistical Analysis Plan: STATISTICAL ANALYSIS (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04707014/SAP_001.pdf
  • Informed Consent Form (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04707014/ICF_002.pdf